CLINICAL TRIAL: NCT07042516
Title: Safety and Efficacy of Asimadoline (TP0052), a Peripherally Restricted Selective Kappa Agonist, for the Treatment of Moderate to Severe Menopausal Symptoms in Midlife Women.
Brief Title: Safety and Efficacy of Asimadoline (TP0052) in Patients With Vasomotor Symptoms (VMS).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tioga Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIOGA VMS-08; IND#: 160,058 (Other: FDA); IRB Tracking Number: 20250414 (Other: WCG IRB)
Record Dates: First submitted 2025-06-19; First posted 2025-06-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Vasomotor Symptoms
Keywords: vasomotor symptoms; VMS; asimadoline; perimenopausal; postmenopausal; hot flashes
MeSH Terms: conditions — Hot Flashes | interventions — asimadoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Asimadoline (Experimental): Asimadoline TP0052 2.5 mg two (2) tablets bid (two on awakening and two before bed), total of four (4) tablets daily (10 mg) for 8 weeks. Post-unblinding 4 weeks of open label administration, TP0052 2.5 mg two (2) tablets bid (two on awakening and two before bed), total of four (4) tablets daily (10 mg) for 4 weeks.
  Interventions: Drug: Asimadoline
- Placebo (Placebo Comparator): Placebo two (2) tablets bid (two on awakening and two before bed), total of four (4) tablets daily for 8 weeks.
  Interventions: Drug: Asimadoline

INTERVENTIONS:
Drug: Asimadoline — Asimadoline TP0052 2.5 mg two (2) tablets bid (two on awakening and two before bed), total of four (4) tablets daily (10 mg) for 8 weeks.
  Other Names: TP0052

SUMMARY:
This Randomized Clinical Trial entitled Safety and Efficacy of a Peripherally Restricted Selective Kappa Agonist for Moderate to Severe Menopausal Symptoms in Midlife Women is a Phase 2a randomized, double-blind, placebo-controlled trial evaluating the safety and efficacy of asimadoline TP0052 for the treatment of moderate to severe menopausal vasomotor symptoms (VMS). The design includes: 2 weeks of daily recording of VMS prior to drug treatment; 8 weeks of double-blind treatment with the peripherally restricted kappa agonist (PRKA), asimadoline TP0052, or placebo; and a safety telephone follow-up post-treatment; after the initial 8-week double-blinded follow-up, all patients undergo treatment with Asimadoline in an open label format for 4 weeks.

ELIGIBILITY:
Inclusion Criteria

* Females aged 40-62 years.
* Untreated patients (either newly diagnosed with VMS or those with a history of VMS but have not been taking drugs that could have an effect on VMS (e.g., SSRIs, SNRIs, gabapentin, pregabalin, clonidine).
* Menopausal OR late perimenopausal according to the following criteria:

Criteria for Menopause:

* Women who have had a bi-lateral oophorectomy (> 6 weeks prior); OR
* Women with a uterus who have had no vaginal bleeding the past 12 months; OR
* Women without a uterus (or women with a uterus who have either a levonorgestrel intrauterine device [LNG IUD] or who have had an endometrial ablation) and who still have one or both ovaries, with follicle stimulating hormone (FSH) level > 40 mIU/mL and estradiol ≤ 50 pg/mL (on at least one of two blood draws two weeks apart);

Criteria for Late Perimenopause:

* Women with a uterus who have had consecutive intervals of amenorrhea of at least 60 days for three or more cycles (i.e., three consecutive episodes of vaginal bleeding separated by 60 or more days between vaginal bleeding episodes).

  • At least 40 moderate to severe VMS per week for each of the 2 screening weeks, as reported on daily VMS diaries.
* Including at least 6 moderate to severe VMS per day on 4 or more days in each of the 2 screening weeks.
* VMS frequency in week 2 cannot drop by more than 50% from the average weekly level reported during week 1.

  * In general good health as determined by medical history, blood pressure, and heart rate.
  * Signed informed consent.

Exclusion Criteria

* • Use of hormone therapy or hormonal contraceptives (with the exception of the LNG IUD) during the 8 weeks before Screening Visit 1. Use of low-dose vaginal estrogen therapies is allowed, with the exception of vaginal creams used >3 times a week.
* Use of non-hormonal medications that can influence VMS during the 4 weeks before Screening Visit 1, including selective serotonin reuptake inhibitors (SSRIs), selective serotonin-norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin, and clonidine.
* Use of marijuana or cannabis-derived products (including THC or CBD in any form other than topical, including smoked, vaporized, or edible) that can affect central thermoregulatory processes, mood and perception of VMS, and potentially have pharmacodynamic interactions with the asimadoline during the 4 weeks before Screening Visit 1 as determined by interview and urine drug test.
* Use of supplements or herbal therapies that can affect VMS including black cohosh, red clover, dong quai, evening primrose oil, maca, ginseng, chasteberry, milk thistle, and phytoestrogens during the 4 weeks before Screening Visit 1.
* Any current severe or unstable medical illness, including the following:

  * Hypertension of stage 2 or greater (systolic blood pressure ≥ 140 or diastolic blood pressure ≥ 90)
  * Resting heart rate >100.
  * Current cancer diagnosis, except non-melanoma skin cancer, or any findings suggestive of or indicating breast malignancy.
  * Current abnormal Pap smear, breast exam, or mammogram.
  * Coronary artery disease, or cerebrovascular disease.
  * Moderate to severe substance use disorder in the previous 12 months; suicide attempt in the previous 36 months, any major depressive episode within the previous 12 months, or lifetime diagnosis of psychosis or bipolar disorder.
* Pregnancy, intending pregnancy, breast feeding.
* Current participation in another drug trial or intervention study.
* Inability or unwillingness to complete the study procedures.

Trial-Specific Exclusion Criteria:

* Known hypersensitivity to asimadoline TP0052.
* Chronic liver or renal disease, or uncontrolled seizure disorder.
* Use of medications or supplements that act as an inhibitor of P-glycoprotein or as a P-glycoprotein substrate during the 4 weeks prior to Screening Visit 1, including cyclosporine, non-topical ketoconazole, verapamil, digoxin, colchicine, sitagliptin).
* Blood test results indicating:

  * Liver function tests: AST ≥2 times upper limit of normal; ALT ≥2 times upper limit of normal; total bilirubin ≥ 1.5 times upper limit of normal
  * Kidney function test: estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m²
  * Blood count: hematocrit <30%.

Ages: 40 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Safety as Assessed by Adverse Events, Clinical Laboratory Parameters, and Vital Signs | baseline to 8 weeks
  Safety will be evaluated based on the incidence and severity of adverse events and changes from baseline in laboratory values and vital signs. Adverse events will be graded using the Common Terminology Criteria for Adverse Events, Version 5.0 (grade 1 = mild; grade 5 = death; higher scores indicate worse outcomes). Liver function tests include alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, alkaline phosphatase, and total bilirubin. Higher values indicate worse liver function. Kidney function will be assessed by estimated glomerular filtration rate (scale: 0 to ≥90 mL/min/1.73 m²; <60 considered abnormal; higher is better). Hematocrit will be monitored (percent; <30% is abnormal; higher is better within normal range). Vital signs include blood pressure, heart rate, respiratory rate, and oral temperature; higher blood pressure and heart rate indicate worse outcomes. A urine pregnancy test (positive or negative) will also be performed.

SECONDARY OUTCOMES:
Change in Frequency of Moderate to Severe Vasomotor Symptoms (VMS) | Baseline to 8 weeks
  The frequency of moderate and severe vasomotor symptoms (VMS) will be measured using participant-completed diaries (paper or electronic) recorded twice daily (morning and evening) from Baseline to Week 8.
  VMS frequency is defined as the number of moderate or severe hot flashes or night sweats reported per day.
  Moderate VMS: sensation of heat with sweating, without disruption of activity. Severe VMS: sensation of heat with sweating that causes cessation of activity or awakening at night.
  The outcome is calculated as the average number of moderate/severe VMS episodes per day, averaged over the 8-week treatment period.
  Due to protocol-defined eligibility criteria, all participants will report at least 40 moderate/severe VMS episodes per week at baseline. During treatment, the minimum possible observed value is 0 episodes/day. There is no fixed upper limit; values of 20-30 episodes/day may occur.
  Higher values indicate worse symptom frequency.
Change in Severity-Weighted Vasomotor Symptom (VMS) Score (Composite Severity Index). | Baseline to 8 weeks
  VMS severity will be assessed using a composite score derived from participant diaries recorded twice daily from Baseline to Week 8.
  Each VMS episode is assigned a severity score:
  Mild = 1 Moderate = 2 Severe = 3
  Daily VMS severity scores are calculated as:
  (# Mild × 1) + (# Moderate × 2) + (# Severe × 3)
  Weekly averages of daily severity scores are computed for each participant. The average across the 8-week treatment period will serve as the outcome measure.
  Due to protocol-defined eligibility criteria, all participants will report ≥40 moderate/severe VMS episodes per week at baseline. During treatment, the minimum possible observed value is 0. There is no fixed upper limit; for example, 10 severe episodes per day would result in a score of 30.
  Higher scores indicate worse symptom severity.

OTHER OUTCOMES:
Exploratory Outcome Measure - Change in VMS (vasomotor symptoms) Bothersomeness Score | Baseline to 8 weeks
  Participant-reported bothersomeness of vasomotor symptoms (VMS) will be assessed using a numeric rating scale completed twice daily (morning and evening) via VMS diaries from Baseline to Week 8.
  Scale: 0 (not bothersome at all) to 10 (extremely bothersome) Minimum = 0 Maximum = 10 Higher scores indicate greater VMS-related bother.
Exploratory Outcome Measure - Change in Sleep Quality Rating | Baseline to 8 weeks
  Sleep quality will be assessed via participant-reported ratings recorded in daily VMS diaries twice daily (morning and evening) from Baseline to Week 8. Participants will indicate the degree to which VMS disrupted their sleep using a 0-10 numeric scale.
  Minimum score: 0 (no disruption to sleep) Maximum score: 10 (extreme disruption to sleep) Higher scores indicate worse sleep quality.
Exploratory Outcome Measure - Change in Menopause-Specific Quality of Life (MENQOL) Score. | Baseline to 8 weeks
  Quality of life will be measured using the MENQOL questionnaire, a validated 29-item scale assessing four domains: vasomotor, psychosocial, physical, and sexual. Participants will complete the MENQOL at baseline and at Week 8.
  Scale range per item: 1 (not at all bothered) to 8 (extremely bothered) Overall score = mean of all item responses Minimum = 1 Maximum = 8 Higher scores indicate worse menopause-related quality of life.
Exploratory Outcome Measure - Change in Female Sexual Function Index (FSFI) Score. | Baseline to 8 weeks
  Sexual functioning will be assessed using the FSFI questionnaire, a validated 19-item instrument covering desire, arousal, lubrication, orgasm, satisfaction, and pain. FSFI will be administered at Baseline and Week 8.
  Scale total range: 2 to 36 Minimum = 2 Maximum = 36 Higher scores indicate better sexual functioning.
Exploratory Outcome Measure - Change in Pain Intensity Rating. | Baseline to 8 weeks
  Pain intensity will be assessed via participant self-report using a numeric rating scale (NRS), recorded at Baseline and Week 8. Participants will rate the severity of pain symptoms potentially associated with menopausal status or treatment effect.
  Minimum score: 0 (no pain) Maximum score: 10 (worst pain imaginable) Higher scores indicate worse pain.
Exploratory Outcome Measure - Change in Follicle Stimulating Hormone (FSH) Level. | Baseline to 8 weeks
  Serum follicle stimulating hormone (FSH) levels will be measured at Baseline and Week 8 to assess hormonal changes related to treatment.
  Units: mIU/mL No fixed minimum or maximum; normal postmenopausal levels typically >40 mIU/mL Directional hypothesis: decreasing FSH may correlate with treatment response.
Exploratory Outcome Measure - Change in Adiponectin Level | Baseline to 8 weeks
  Serum adiponectin will be measured at Baseline and Week 8 to explore its correlation with VMS treatment response.
  Units: μg/mL Directional hypothesis: modulation may indicate metabolic effects of treatment Higher or lower values will be analyzed for association with response.
Exploratory Outcome Measure - Change in C-Reactive Protein (CRP) Level | Baseline to 8 weeks
  High-sensitivity CRP (hsCRP) will be measured at Baseline and Week 8 as a marker of systemic inflammation.
  Units: mg/L Typical reference range: <3.0 mg/L Changes will be evaluated for correlation with treatment response.
Exploratory Outcome Measure - Change in Leptin Level. | Baseline to 8 weeks
  Serum leptin will be measured at Baseline and Week 8 to evaluate metabolic and hypothalamic correlates of treatment effect.
  Units: ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dunlop - Principal Investigator, MD, Principal Investigator — Emory University; Sergey Sikora, VP of Clinical Affairs, PhD, Study Chair — Tioga Pharmaceuticals
Locations (1):
- Department of Gynecology & Obstetrics, Emory University School of Medicine, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Description:
  De-identified individual participant data (IPD) will be made available to qualified researchers upon reasonable request. Access will be granted following approval of a research proposal and execution of a data-sharing agreement. Data will be shared through a secure platform to ensure confidentiality and compliance with applicable regulations. The shared data may include clinical study reports, anonymized participant-level datasets, and relevant supporting documentation.
  Time Frame:
  Data will be available upon publication of the primary study results and for a period of 5 years thereafter.
  Access Criteria:
  Researchers must submit a detailed proposal outlining the intended use of the data. Proposals will be reviewed by an independent data-sharing committee. Approved researchers must adhere to ethical and security guidelines, ensuring proper data use in compliance with applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] National Institutes of Health. National Institutes of Health State-of-the-Science Conference statement: management of menopause-related symptoms. Ann Intern Med. 2005 Jun 21;142(12 Pt 1):1003-13. Epub 2005 May 27. No abstract available. PMID 15968015
- [Background] Anderson GL, Limacher M, Assaf AR, Bassford T, Beresford SA, Black H, Bonds D, Brunner R, Brzyski R, Caan B, Chlebowski R, Curb D, Gass M, Hays J, Heiss G, Hendrix S, Howard BV, Hsia J, Hubbell A, Jackson R, Johnson KC, Judd H, Kotchen JM, Kuller L, LaCroix AZ, Lane D, Langer RD, Lasser N, Lewis CE, Manson J, Margolis K, Ockene J, O'Sullivan MJ, Phillips L, Prentice RL, Ritenbaugh C, Robbins J, Rossouw JE, Sarto G, Stefanick ML, Van Horn L, Wactawski-Wende J, Wallace R, Wassertheil-Smoller S; Women's Health Initiative Steering Committee. Effects of conjugated equine estrogen in postmenopausal women with hysterectomy: the Women's Health Initiative randomized controlled trial. JAMA. 2004 Apr 14;291(14):1701-12. doi: 10.1001/jama.291.14.1701. PMID 15082697
- [Background] Avis NE, Stellato R, Crawford S, Bromberger J, Ganz P, Cain V, Kagawa-Singer M. Is there a menopausal syndrome? Menopausal status and symptoms across racial/ethnic groups. Soc Sci Med. 2001 Feb;52(3):345-56. doi: 10.1016/s0277-9536(00)00147-7. PMID 11330770
- [Background] Appling S, Paez K, Allen J. Ethnicity and vasomotor symptoms in postmenopausal women. J Womens Health (Larchmt). 2007 Oct;16(8):1130-8. doi: 10.1089/jwh.2006.0033. PMID 17937565
- [Background] Freeman EW, Sherif K. Prevalence of hot flushes and night sweats around the world: a systematic review. Climacteric. 2007 Jun;10(3):197-214. doi: 10.1080/13697130601181486. PMID 17487647
- [Background] 35. NCT02475447, Safety, Pharmacokinetics and Preliminary Efficacy of Asimadoline in Pruritus Associated With Atopic Dermatitis. 2017, Tioga Pharmaceuticals: https://clinicaltrials.gov.
- [Background] Mangel AW, Hicks GA. Asimadoline and its potential for the treatment of diarrhea-predominant irritable bowel syndrome: a review. Clin Exp Gastroenterol. 2012;5:1-10. doi: 10.2147/CEG.S23274. Epub 2012 Jan 12. PMID 22346361
- [Background] Wakabayashi Y, Nakada T, Murata K, Ohkura S, Mogi K, Navarro VM, Clifton DK, Mori Y, Tsukamura H, Maeda K, Steiner RA, Okamura H. Neurokinin B and dynorphin A in kisspeptin neurons of the arcuate nucleus participate in generation of periodic oscillation of neural activity driving pulsatile gonadotropin-releasing hormone secretion in the goat. J Neurosci. 2010 Feb 24;30(8):3124-32. doi: 10.1523/JNEUROSCI.5848-09.2010. PMID 20181609
- [Background] Trower M, Anderson RA, Ballantyne E, Joffe H, Kerr M, Pawsey S. Effects of NT-814, a dual neurokinin 1 and 3 receptor antagonist, on vasomotor symptoms in postmenopausal women: a placebo-controlled, randomized trial. Menopause. 2020 May;27(5):498-505. doi: 10.1097/GME.0000000000001500. PMID 32068688
- [Background] Lederman S, Ottery FD, Cano A, Santoro N, Shapiro M, Stute P, Thurston RC, English M, Franklin C, Lee M, Neal-Perry G. Fezolinetant for treatment of moderate-to-severe vasomotor symptoms associated with menopause (SKYLIGHT 1): a phase 3 randomised controlled study. Lancet. 2023 Apr 1;401(10382):1091-1102. doi: 10.1016/S0140-6736(23)00085-5. Epub 2023 Mar 13. PMID 36924778
- [Background] Johnson KA, Martin N, Nappi RE, Neal-Perry G, Shapiro M, Stute P, Thurston RC, Wolfman W, English M, Franklin C, Lee M, Santoro N. Efficacy and Safety of Fezolinetant in Moderate to Severe Vasomotor Symptoms Associated With Menopause: A Phase 3 RCT. J Clin Endocrinol Metab. 2023 Jul 14;108(8):1981-1997. doi: 10.1210/clinem/dgad058. PMID 36734148
- [Background] Prague JK, Roberts RE, Comninos AN, Clarke S, Jayasena CN, Nash Z, Doyle C, Papadopoulou DA, Bloom SR, Mohideen P, Panay N, Hunter MS, Veldhuis JD, Webber LC, Huson L, Dhillo WS. Neurokinin 3 receptor antagonism as a novel treatment for menopausal hot flushes: a phase 2, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 6;389(10081):1809-1820. doi: 10.1016/S0140-6736(17)30823-1. Epub 2017 Apr 3. PMID 28385352
- [Background] Rance NE, Dacks PA, Mittelman-Smith MA, Romanovsky AA, Krajewski-Hall SJ. Modulation of body temperature and LH secretion by hypothalamic KNDy (kisspeptin, neurokinin B and dynorphin) neurons: a novel hypothesis on the mechanism of hot flushes. Front Neuroendocrinol. 2013 Aug;34(3):211-27. doi: 10.1016/j.yfrne.2013.07.003. Epub 2013 Jul 17. PMID 23872331
- [Background] Oakley AE, Steiner RA, Chavkin C, Clifton DK, Ferrara LK, Reed SD. kappa Agonists as a novel therapy for menopausal hot flashes. Menopause. 2015 Dec;22(12):1328-34. doi: 10.1097/GME.0000000000000476. PMID 25988798
- [Background] 26. FDA, BRISDELLE (paroxetine mesylate) NDA 204516 Approval Letter. U.S. Food and Drug Administration, Center for Drug Evaluation and Research, 2013.
- [Background] Joffe H, Guthrie KA, LaCroix AZ, Reed SD, Ensrud KE, Manson JE, Newton KM, Freeman EW, Anderson GL, Larson JC, Hunt J, Shifren J, Rexrode KM, Caan B, Sternfeld B, Carpenter JS, Cohen L. Low-dose estradiol and the serotonin-norepinephrine reuptake inhibitor venlafaxine for vasomotor symptoms: a randomized clinical trial. JAMA Intern Med. 2014 Jul;174(7):1058-66. doi: 10.1001/jamainternmed.2014.1891. PMID 24861828
- [Background] Freeman EW, Guthrie KA, Caan B, Sternfeld B, Cohen LS, Joffe H, Carpenter JS, Anderson GL, Larson JC, Ensrud KE, Reed SD, Newton KM, Sherman S, Sammel MD, LaCroix AZ. Efficacy of escitalopram for hot flashes in healthy menopausal women: a randomized controlled trial. JAMA. 2011 Jan 19;305(3):267-74. doi: 10.1001/jama.2010.2016. PMID 21245182
- [Background] Barton DL, Loprinzi CL, Novotny P, Shanafelt T, Sloan J, Wahner-Roedler D, Rummans TA, Christensen B, Dakhill SR, Martin LS. Pilot evaluation of citalopram for the relief of hot flashes. J Support Oncol. 2003 May-Jun;1(1):47-51. PMID 15352642
- [Background] Loprinzi CL, Sloan JA, Perez EA, Quella SK, Stella PJ, Mailliard JA, Halyard MY, Pruthi S, Novotny PJ, Rummans TA. Phase III evaluation of fluoxetine for treatment of hot flashes. J Clin Oncol. 2002 Mar 15;20(6):1578-83. doi: 10.1200/JCO.2002.20.6.1578. PMID 11896107
- [Background] Rapkin AJ. Vasomotor symptoms in menopause: physiologic condition and central nervous system approaches to treatment. Am J Obstet Gynecol. 2007 Feb;196(2):97-106. doi: 10.1016/j.ajog.2006.05.056. PMID 17306645
- [Background] Suvanto-Luukkonen E, Koivunen R, Sundstrom H, Bloigu R, Karjalainen E, Haiva-Mallinen L, Tapanainen JS. Citalopram and fluoxetine in the treatment of postmenopausal symptoms: a prospective, randomized, 9-month, placebo-controlled, double-blind study. Menopause. 2005 Jan-Feb;12(1):18-26. doi: 10.1097/00042192-200512010-00006. PMID 15668596
- [Background] Grady D, Cohen B, Tice J, Kristof M, Olyaie A, Sawaya GF. Ineffectiveness of sertraline for treatment of menopausal hot flushes: a randomized controlled trial. Obstet Gynecol. 2007 Apr;109(4):823-30. doi: 10.1097/01.AOG.0000258278.73505.fa. PMID 17400842
- [Background] Stearns V, Slack R, Greep N, Henry-Tilman R, Osborne M, Bunnell C, Ullmer L, Gallagher A, Cullen J, Gehan E, Hayes DF, Isaacs C. Paroxetine is an effective treatment for hot flashes: results from a prospective randomized clinical trial. J Clin Oncol. 2005 Oct 1;23(28):6919-30. doi: 10.1200/JCO.2005.10.081. PMID 16192581
- [Background] Loprinzi CL, Kugler JW, Sloan JA, Mailliard JA, LaVasseur BI, Barton DL, Novotny PJ, Dakhil SR, Rodger K, Rummans TA, Christensen BJ. Venlafaxine in management of hot flashes in survivors of breast cancer: a randomised controlled trial. Lancet. 2000 Dec 16;356(9247):2059-63. doi: 10.1016/S0140-6736(00)03403-6. PMID 11145492
- [Background] Shaver JL. Beyond hormonal therapies in menopause. Exp Gerontol. 1994 May-Aug;29(3-4):469-76. doi: 10.1016/0531-5565(94)90027-2. PMID 7925765
- [Background] Stearns V, Ullmer L, Lopez JF, Smith Y, Isaacs C, Hayes D. Hot flushes. Lancet. 2002 Dec 7;360(9348):1851-61. doi: 10.1016/s0140-6736(02)11774-0. PMID 12480376
- [Background] Freedman RR, Woodward S, Sabharwal SC. Alpha 2-adrenergic mechanism in menopausal hot flushes. Obstet Gynecol. 1990 Oct;76(4):573-8. PMID 2170883
- [Background] 13. Freedman, R. and S. Woodward, Elevated α2-adrenergic responsiveness in menopausal hot flushes: pharmacologic and biochemical studies. Thermoregulation: the pathophysiological basis of clinical disorders. Basel: Karger, 1992: p. 6-9.
- [Background] Bruck K, Zeisberger E. Adaptive changes in thermoregulation and their neuropharmacological basis. Pharmacol Ther. 1987;35(1-2):163-215. doi: 10.1016/0163-7258(87)90106-9. PMID 3321099
- [Background] 11. Freedman, R.R. Pathophysiology and treatment of menopausal VMS. in Seminars in reproductive medicine. 2005. Copyright© 2005 by Thieme Medical Publishers, Inc., 333 Seventh Avenue, New York, NY 10001, USA.
- [Background] 10. FDA, VEOZAH™ (fezolinetant) tablets, for oral use: NDA 216578 Approval Letter. U.S. Food and Drug Administration, Center for Drug Evaluation and Research, 2023.
- [Background] Simon JA, Portman DJ, Kaunitz AM, Mekonnen H, Kazempour K, Bhaskar S, Lippman J. Low-dose paroxetine 7.5 mg for menopausal vasomotor symptoms: two randomized controlled trials. Menopause. 2013 Oct;20(10):1027-35. doi: 10.1097/GME.0b013e3182a66aa7. PMID 24045678
- [Background] Carroll DG. Nonhormonal therapies for hot flashes in menopause. Am Fam Physician. 2006 Feb 1;73(3):457-64. PMID 16477892
- [Background] Geller SE, Studee L. Botanical and dietary supplements for mood and anxiety in menopausal women. Menopause. 2007 May-Jun;14(3 Pt 1):541-9. doi: 10.1097/01.gme.0000236934.43701.c5. PMID 17194961
- [Background] Newton KM, Reed SD, LaCroix AZ, Grothaus LC, Ehrlich K, Guiltinan J. Treatment of vasomotor symptoms of menopause with black cohosh, multibotanicals, soy, hormone therapy, or placebo: a randomized trial. Ann Intern Med. 2006 Dec 19;145(12):869-79. doi: 10.7326/0003-4819-145-12-200612190-00003. PMID 17179056
- [Background] Tremblay A, Sheeran L, Aranda SK. Psychoeducational interventions to alleviate hot flashes: a systematic review. Menopause. 2008 Jan-Feb;15(1):193-202. doi: 10.1097/gme.0b013e31805c08dc. PMID 17589375
- [Background] Buist DS, Newton KM, Miglioretti DL, Beverly K, Connelly MT, Andrade S, Hartsfield CL, Wei F, Chan KA, Kessler L. Hormone therapy prescribing patterns in the United States. Obstet Gynecol. 2004 Nov;104(5 Pt 1):1042-50. doi: 10.1097/01.AOG.0000143826.38439.af. PMID 15516400
- [Background] Haas JS, Kaplan CP, Gerstenberger EP, Kerlikowske K. Changes in the use of postmenopausal hormone therapy after the publication of clinical trial results. Ann Intern Med. 2004 Feb 3;140(3):184-8. doi: 10.7326/0003-4819-140-3-200402030-00009. PMID 14757616
- [Background] Grady D, Ettinger B, Tosteson AN, Pressman A, Macer JL. Predictors of difficulty when discontinuing postmenopausal hormone therapy. Obstet Gynecol. 2003 Dec;102(6):1233-9. doi: 10.1016/j.obstetgynecol.2003.09.025. PMID 14662209
- [Background] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397